CLINICAL TRIAL: NCT07133828
Title: A Phase 1, Randomized, Blinded, Placebo-Controlled, Single- and Multiple-Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of BIIB142 in Healthy Adults
Brief Title: A Study to Learn About the Safety of BIIB142 and How it is Processed in the Body of Healthy Adult Participants Aged 18 to 55 Years Old
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 300HV101
Record Dates: First submitted 2025-08-14; First posted 2025-08-21 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Part A [Single Ascending Dose (SAD)]: BIIB142Cohort 1A (Experimental): Participants will receive Dose A of BIIB142 or a matching placebo on Day 1 in a fasted state.
  Interventions: Drug: BIIB142; Drug: BIIB142-Matching Placebo
- Part A (SAD): BIIB142 Cohort 2A (Experimental): Participants will receive Dose B of BIIB142 or a matching placebo on Day 1 in a fasted state.
  Interventions: Drug: BIIB142; Drug: BIIB142-Matching Placebo
- Part A (SAD): BIIB142 Cohort 3A (Experimental): Participants will receive Dose C of BIIB142 or a matching placebo on Day 1 in a fasted state.
  Interventions: Drug: BIIB142; Drug: BIIB142-Matching Placebo
- Part A (SAD): BIIB142 Cohort 4A (Experimental): Participants will receive Dose D of BIIB142 or a matching placebo on Day 1 in a fasted state.
  Interventions: Drug: BIIB142; Drug: BIIB142-Matching Placebo
- Part A (SAD): BIIB142 Cohort 5A (Experimental): Participants will receive Dose E of BIIB142 or a matching placebo on Day 1 in a fasted state.
  Interventions: Drug: BIIB142; Drug: BIIB142-Matching Placebo
- Part A (SAD): BIIB142 Cohort 6A (Experimental): Participants will receive BIIB142 on Day 1 in the fasted followed by fed state in the first sequence, and vice versa in the second sequence. A washout period of 14 days will be maintained between both the sequences. Dose will be determined based on emerging PK data.
  Interventions: Drug: BIIB142
- Part B [Multiple Ascending Dose (MAD)]: BIIB142 Cohort 1B (Experimental): Participants will receive Dose A of BIIB142 or a matching placebo administered orally once daily for 14 days in a fasted state.
  Interventions: Drug: BIIB142; Drug: BIIB142-Matching Placebo
- Part B (MAD): BIIB142 Cohort 2B (Experimental): Participants will receive Dose F of BIIB142 or a matching placebo administered orally once daily for 14 days in a fasted state.
  Interventions: Drug: BIIB142; Drug: BIIB142-Matching Placebo
- Part B (MAD): BIIB142 Cohort 3B (Experimental): Participants will receive Dose D of BIIB142 or a matching placebo administered orally once daily for 14 days in a fasted state.
  Interventions: Drug: BIIB142; Drug: BIIB142-Matching Placebo

INTERVENTIONS:
Drug: BIIB142 — Administered Orally
Drug: BIIB142-Matching Placebo — Administered Orally
  Arms: Part A (SAD): BIIB142 Cohort 2A; Part A (SAD): BIIB142 Cohort 3A; Part A (SAD): BIIB142 Cohort 4A; Part A (SAD): BIIB142 Cohort 5A; Part A [Single Ascending Dose (SAD)]: BIIB142Cohort 1A; Part B (MAD): BIIB142 Cohort 2B; Part B (MAD): BIIB142 Cohort 3B; Part B [Multiple Ascending Dose (MAD)]: BIIB142 Cohort 1B

SUMMARY:
In this study, researchers will learn more about the safety of BIIB142 and how it is processed in the body. This is the first time that researchers will learn about BIIB142 and how it affects people.

The main question researchers want to answer in this study is:

• How many participants have adverse events (AEs) and serious adverse events (SAEs)?

An AE is a health problem that may or may not be caused by a drug during the study. An AE is considered serious when it results in death, is life-threatening, causes lasting problems, or requires hospital care.

Researchers will also learn more about:

• How the body processes BIIB142

This is a "dose escalation study." This is a study in which increasing amounts of the study drug are given to different groups of participants. This is done until researchers find the highest dose that does not cause harmful effects.

First, participants will be screened to check if they can join the study. The screening period will be up to 28 days. This study will be split into 2 parts - Part A and Part B.

During Part A:

* Participants will be randomly placed into 1 of 6 groups to receive a single dose of either BIIB142 or a placebo. A placebo looks like the study drug but contains no real medicine.
* Participants in Groups 1 through 5 will take either BIIB142 or the placebo without food. Participants in Group 6 will take 2 doses of their assigned treatment - once with food and once without food.
* Neither the researchers nor the participants will know if the participants will receive BIIB142 or the placebo.
* Participants will stay at their study research center for 5 days. They will return for another 4 visits. Each participant in Part A will be in the study for up to 58 days.

During Part B:

* Participants will be randomly placed into 1 of 3 groups to receive BIIB142 or the placebo. In Part B, participants will take BIIB142 or the placebo once a day for 14 days.
* Neither the researchers nor the participants will know if the participants will receive BIIB142 or the placebo.
* Participants will stay at their study research center for 16 days. They will return for another 4 visits. Each participant in Part B will be in the study for up to 58 days.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and tolerability of single and multiple ascending oral doses of BIIB142 in healthy adult participants.

The secondary objective of this study is to evaluate the pharmacokinetics (PK) profile of single and multiple ascending oral doses of BIIB142 in healthy adult participants.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a body mass index between 18 and 32 kilograms per square meter (kg/m^2), inclusive, at screening.
* Weight ≥ 50 kilograms (kg) at screening.
* Negative polymerase chain reaction (PCR) test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) at Check-in prior to randomization.
* Must be in good health as determined by the Investigator.

Key Exclusion Criteria:

* History of any clinically significant cardiac, endocrine, gastrointestinal, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, or renal disease, or other major disease, as determined by the Investigator.
* History of severe allergic or anaphylactic reactions
* History of or ongoing malignant disease (with limited exceptions)
* Systolic blood pressure >150 millimeters of mercury (mmHg) or <90 mmHg.
* Clinically significant (as determined by the Investigator) electrocardiogram (ECG) abnormalities.
* History of or positive test for human immunodeficiency virus (HIV).
* Chronic, recurrent, or serious infection within 90 days prior to Screening.
* Symptoms of bacterial, fungal, or viral infection within 14 days prior to Screening.
* Any live or attenuated immunization within 14 days prior to Screening.
* Use of prescription medications, over-the-counter medications that alter hepatic or renal clearance, or nutraceuticals within 28 days prior to Check-in.
* MAD Cohorts only: Suicidal ideation with some intent to act within 6 months prior to the start of Screening or history of suicidal behavior within one year prior to Screening.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2026-08-06 (Estimated); Study Completion 2026-08-06 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Part A (SAD): Up to Day 15; Part B (MAD): Up to Day 29
Number of Participants with Clinical Laboratory Abnormalities | Part A (SAD): Up to Day 15; Part B (MAD): Up to Day 29
Number of Participants with Potentially Clinically Relevant Abnormalities in Vital Sign Parameters | Part A (SAD): Up to Day 15; Part B (MAD): Up to Day 29
Number of Participants With Change From Baseline in Columbia Suicide Severity Rating Scale (C-SSRS) Score | Part B (MAD): Up to Day 29
Number of Participants With Potentially Clinically Relevant Abnormalities in 12-lead Electrocardiogram (ECG) Parameters | Part A (SAD): Up to Day 15; Part B (MAD): Up to Day 29

SECONDARY OUTCOMES:
Plasma Concentration of BIIB142 | Pre-dose and at multiple timepoints post-dose [Part A (SAD): Up to Day 15; Part B (MAD): Up to Day 29]
Area Under the Concentration-Time Curve (AUC) of BIIB142 | Pre-dose and at multiple timepoints post-dose [Part A (SAD): Up to Day 15; Part B (MAD): Up to Day 29]
Maximum Observed Concentration (Cmax) of BIIB142 | Pre-dose and at multiple timepoints post-dose [Part A (SAD): Up to Day 15; Part B (MAD): Up to Day 29]
Time to Maximum Observed Concentration (Tmax) of BIIB142 | Pre-dose and at multiple timepoints post-dose [Part A (SAD): Up to Day 15; Part B (MAD): Up to Day 29]
Apparent Clearance (CL/F) of BIIB142 | Pre-dose and at multiple timepoints post-dose [Part A (SAD): Up to Day 15; Part B (MAD): Up to Day 29]
Apparent Volume of Distribution (Vz/F) of BIIB142 | Pre-dose and at multiple timepoints post-dose [Part A (SAD): Up to Day 15; Part B (MAD): Up to Day 29]
Elimination Half-Life (t1/2) of BIIB142 | Pre-dose and at multiple timepoints post-dose [Part A (SAD): Up to Day 15; Part B (MAD): Up to Day 29]

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, LP, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/